CLINICAL TRIAL: NCT02129985
Title: Effect of Short-term Intensive Insulin Sequential Exenatide Therapy on Beta Cell Function and Glycaemic Control in Patients With Newly Diagnosed Type 2 Diabetes :a Multicenter Prospective Randomized Control Study
Brief Title: Effect on Beta Cell Function and Glycaemic Control After Insulin and Exenatide Sequential Therapy
Acronym: T2DMRS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: xiaolong zhao (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); The third people's Hospital Affiliated to Shanghai Jiao Tong University (Unknown); Second Affiliated Hospital of Soochow University (Other); The First Hospital of Guiyang Medical college (Unknown); Fuling Central Hospital of Chongqing City (Other); Taizhou Hospital (Other); Shanghai Pudong New Area Gongli Hospital (Other)
Responsible Party: Sponsor-Investigator, xiaolong zhao, Endocrinology department, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS2014-005
Record Dates: First submitted 2014-04-10; First posted 2014-05-02 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-04

CONDITIONS: Type 2 Diabetes
Keywords: the newly onset type 2 diabetes; short-term insulin treatment; exenatide sequential therapy; beta cell function; glycaemic remission
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Experimental): patients were all received a short-term intensive insulin therapy,then randomised to Exenatide group(10 ug two times a day for three months)
  Interventions: Drug: Exenatide
- Metformin (Active Comparator): patients were all received a short-term intensive insulin therapy,then randomised to metformin group(850mg two times a day for three months)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Exenatide — Exenatide (10 ug/bid for 3 months)
  Other Names: GLP-1 receptor agonist
  Arms: Exenatide
Drug: Metformin — Metformin 850 mg/bid for 3 months
  Other Names: Glucophage
  Arms: Metformin

SUMMARY:
Whether GLP-1 receptor agonists sequential therapy in newly diagnosed type 2 diabetic patients can further improve glycemic control, diabetes remission rate and β-cell function after the short-term insulin intensive therapy.

DETAILED DESCRIPTION:
The UK Prospective Diabetes Study has shown that β-cell function progressively deteriorates over time in people with type 2 diabetes mellitus,irrespective of lifestyle and existing pharmacological interventions. The progressive nature of type 2 diabetes is one of the major challenges in the treatment of affected patients, and agents that could alter the natural history of this condition would add greatly to current treatment approaches.Short-term intensive insulin therapy of newly diagnosed type 2 diabetes has been proved improving beta-cell function and usually leading to a temporary remission time,but the remission rate in a year is only about 50%. The effect of GLP-1 receptor agonists on beta-cells is stimulation of glucose-dependent insulin release, followed by enhancement of insulin biosynthesis. It is stimulating beta-cell proliferation, induction of islet neogenesis, and inhibition of ß-cell apoptosis. Exenatide is an GLP-1 receptor agonist. Exenatide exerts direct effects on β-cell, which indicates that may contribute to delay disease progression. However, no study has evaluated effect of short-term intensive insulin sequential exenatide therapy model on β-cell function and glycemic remission rate in newly diagnosed type 2 diabetic patients. Our hypotheses is whether GLP-1 receptor agonists sequential therapy in newly diagnosed type 2 diabetic patients can further improve glycemic control, diabetes remission rate and β-cell function after the short-term insulin intensive therapy.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed type 2 diabetes without drug treatment
* 25-70 years old age
* Fasting glucose between 7.0-16.7mmol / L
* BMI at 20 ~ 35 kg/m2 and stable for at least 3 month(weight fluctuations within three months does not exceed 10%)
* females who have no plan of pregnancy during the study

Exclusion Criteria:

* acute or chronic complications of diabetes
* myocardial infarction or cerebrovascular events within three months
* serious gastrointestinal diseases
* other serious concomitant diseases
* liver or kidney dysfunction:Transaminase (ALT and AST) greater than 3 times the upper limit of the normal range or creatinine levels greater than 133μmol / L
* GAD antibodies positive
* history of pancreatitis or pancreatic cancer;
* pregnant or breastfeeding women.
* severe hypertension (blood pressure> 180/110mmhg)
* using corticosteroids, immunosuppressants and cytotoxic therapy.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-06 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
time to glycaemic remission | up to 1 year
  time of glycaemic remission at 1 year after exenatide sequential therapy followed by a short-term insulin intensive treatment
remission rate of type 2 diabetes at a year. | up to 1 year
  remission rate of type 2 diabetes after short-term intensive insulin and exenatide sequencial therapy

SECONDARY OUTCOMES:
the beta cell function change | 1 year
  the beta cell function change expressed by the ratio of proinsulin to insulin in fasting state and HOMA beta,the ratio of Glucose change to insulin change between at 30min and 0min time point of OGTT

OTHER OUTCOMES:
HbA1C level at every 3 months during the whole study | 1 year
  HbA1C level at every 3 months during the whole study
mean glucose level during the follow without drug intervention | 1 year
  mean glucose level during the follow without drug intervention
number of hypoglycemia and severe hypoglycemia during the study | up to 1 year
  number of hypoglycemia and severe hypoglycemia during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaolong Zhao, Jingan, Shanghai Municipality, China